CLINICAL TRIAL: NCT03139903
Title: The Primordial Dwarfisms: Diagnosis, Identification of the Molecular Basis of Seckel Syndrome and Microcephalic Osteodysplastic Primordial Dwarfism Type II (MOPDII).
Brief Title: The Primordial Dwarfisms: Diagnosis, Identification of the Molecular Basis of Seckel Syndrome and Microcephalic Osteodysplastic Primordial Dwarfism Type II
Acronym: NANPIM
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: P081256
Record Dates: First submitted 2017-03-23; First posted 2017-05-04 (Actual); Last update posted 2017-11-20 (Actual); Status verified 2017-11

CONDITIONS: Microcephalic Osteodysplastic Primordial Dwarfism Type II; Seckel Syndrome
Keywords: Seckel Syndrome; Microcephalic Osteodysplastic Primordial Dwarfism Type II
MeSH Terms: conditions — Microcephalic Osteodysplastic Primordial Dwarfism, Type II; Seckel syndrome 1

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study si to define morphological and epidemiological parameters and identify new symptoms in French patients with Seckel syndrome (SCKL) or microcephalic osteodysplastic primordial dwarfism type II (MOPDII).

DETAILED DESCRIPTION:
Multicentre study, aiming to determine morphological and epidemiological parameters and identify new symptoms in French patients with SCKL or MOPDII.

At pre-inclusion visit: Realization of the photographs of: the face, entire body and the extremities (hands and feet) that will be serve for the collegiate decision of the inclusion or not of patients.

Patients are seen at inclusion V1 , a second visit V2 at 6-10 months after V1 and an annual follow-up visit.

At inclusion:

* Full Clinical Examination, specialized consultations (Otorhinolaryngology, stomatology, orthopedics, ophthalmology)
* Results of x-ray examinations and biological tests
* Assessment of the patients competencies and initiation of appropriate care ( orthophony and psychomotricity...)
* Assessment of intelligence and cognitive ability according the WISC-IV scale
* Blood testing for diagnosis and research.

Visit 2:

* Full Clinical Examination
* Cerebral angiography-MRI for all patients
* Programming a neurosurgery / neurovascular consultation based on MRI results
* Immuno-hematology and hepato-gastroenterology consultation if anomaly during the visit V1

Annual follow-up visit:

* Assessment of the complications of the disease and its clinical care
* Full clinical examination
* Skeletal x-ray and systematic orthopedic consultation
* Blood Check
* Prescription of tests if necessary depending to the complications identified of the disease
* Reevaluation of the care according to the detected symptoms

ELIGIBILITY:
Inclusion Criteria:

Patients aged from 2 months to 50 years must present all of the following criteria:

* Symmetrical intrauterine growth restriction (IUGR) < - 2 DS, Birth size <-2 DS and Cranial perimeter of birth <-2 DS
* Postnatal growth restriction (size <-4DS)
* Microcephaly <-4DS
* Clinical Diagnosis of Seckel Syndrome or Microcephalic osteodysplastic primordial dwarfism type II (MOPDII) by a geneticist
* Having given free and informed consent

Exclusion Criteria:

* Refutation of the diagnosis
* Parents' refusal to participate in genetic studies once the diagnosis of SCKL or MOPDII has been establish for the patient (major or minor)
* Allergy to gadolinium, contraindicating the realization of an Angio-MRI
* Absence of affiliation to a social security scheme or Universal Health Coverage.

Min Age: 2 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Primordial Dwarfisms have been followed by network geneticists for which there is no systematic and homogeneous collection of biological, radiological and clinical data
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2010-07-28 (Actual); Primary Completion 2013-07-16 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
to visualize any vascular abnormalities according the cerebral angiography-MRI | 10 months

SECONDARY OUTCOMES:
Assessment of intelligence and cognitive ability according the Wechsler Intelligence Scale for Children (WISC-IV) | 2 days
Measurement of visual acuity | 2 days

CONTACTS AND LOCATIONS:
Overall Officials: CORMIER-DAIRE Valérie, PhD, Principal Investigator — Medical Genetics Department and INSERM U781, Necker-Enfants Malades Hospital, 75743 Paris, France
Locations (1):
- Medical Genetics Department and INSERM U781, Necker-Enfants Malades Hospital, Paris, France